CLINICAL TRIAL: NCT07217106
Title: A Retrospective Assessment of Accelerated Guideline-Directed Medical Therapy for Heart Failure
Brief Title: A Study of Accelerated Guideline-Directed Medical Therapy for Heart Failure
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BUS36
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
Keywords: Medical therapy; Implementation; Cardiac remodeling
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- GDMT Clinic: Patients with HF with an abnormal ejection fraction (EF) who were referred to the GDMT clinic and underwent rapid guideline-recommended medication titration.
- Usual Care (RPRD): Patients from the MGH RPRD receiving care since the 2022 United States HF guideline update who were matched in a 2:1 fashion to GDMT clinic patients. Matching was based on age, sex, race, duration of HF, ischemic heart disease, diabetes mellitus, atrial fibrillation and baseline EF.

SUMMARY:
The aim of the study was to evaluate the efficacy and safety of a Guideline-Directed Medical Therapy (GDMT) clinic within a general cardiology practice relative to usual care. This study analyzed data from patients with heart failure (HF) who were referred to the GDMT clinic at Massachusetts General Hospital (MGH). For the comparator arm, patients in the GDMT clinic were matched to data of patients contained within in the MGH Research Patient Data Repository (RPDR).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of HF, including new onset disease
* Established cardiovascular follow up at the hospital
* Received sub-optimal medical care defined as <50% target doses of GDMT agents
* Left ventricular ejection fraction (LVEF) <50%

Exclusion criteria:

* Planned referral to the Advanced HF program
* Decompensated HF
* End-stage kidney disease

  o glomerular filtration rate (GFR) <15 mL/min/1.73m^2 or on renal replacement therapy
* Untreated severe valvular heart disease
* Advanced HF

  * Inotropic support
  * Transplant or mechanical circulatory support (MCS) planned
  * Enrolled in hospice or palliative care
* Life expectancy <12 months due to non-cardiovascular (CV) disease
* Pericardial constriction
* Hypertrophic cardiomyopathy
* Unwillingness or inability to take GDMT
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients Receiving all Four Class I GDMT Drugs at Final Visit of Follow-up | Up to approximately 16 weeks
  Class I GDMT drugs included angiotensin receptor/neprilysin inhibitor (ARNI), evidence-based beta blocker (eBBB), mineralocorticoid receptor antagonist (MRA), sodium-glucose co-transporter-2 inhibitor (SGLT2i) or renin angiotensin system inhibitor (RASi), eBBB, MRA, SGLT2i.

SECONDARY OUTCOMES:
Number Patients Receiving 50% or More of the Target Dose of Four Class I GDMT Drugs at Final Visit of Follow-up | Up to approximately 16 weeks
Number of Patients on a Higher Number of Therapies at Final Visit of Follow-up Compared to Baseline | Baseline and up to approximately 16 weeks
Change From Baseline in New York Heart Association (NYHA) Classification | Baseline and up to approximately 16 weeks
  The NYHA classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity:
  Class I - No limitation of physical activity. Ordinary physical activity does not cause symptoms of HF.
  Class II - Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in symptoms of HF.
  Class III - Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes symptoms of HF.
  Class IV - Unable to carry out any physical activity without symptoms of HF, or symptoms of HF at rest.
Change From Baseline in N-terminal pro B-type Natriuretic Peptide (NT-proBNP) Concentration | Baseline and up to approximately 16 weeks
Change From Baseline in Echocardiography Measurement: LVEF | Baseline and up to approximately 16 weeks
Change From Baseline in Echocardiography Measurement: Left Ventricular End-Diastolic Volume Index (LVEDVi) | Baseline and up to approximately 16 weeks
Change From Baseline in Echocardiography Measurement: Left Ventricular End-Systolic Volume Index (LVESVi) | Baseline and up to approximately 16 weeks
Change From Baseline in Echocardiography Measurement: Left Atrial Volume Index (LAVi) | Baseline and up to approximately 16 weeks
Change From Baseline in Echocardiography Measurement: Left Ventricular Mass Index (LVMi) | Baseline and up to approximately 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States